CLINICAL TRIAL: NCT01777945
Title: Program for Assessment of Capecitabine (Xeloda) Plus Docetaxel First-line Therapies in HER2-negative Metastatic Breast Cancer (XEBRA Study)
Brief Title: XEBRA Study: An Observational Study of Xeloda (Capecitabine) in Combination With Docetaxel in First Line in Participants With HER2-Negative Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28505
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Receiving Capecitabine/Docetaxel: Participants received capecitabine and docetaxel according to individualized physician-prescribed regimens.
  Interventions: Drug: capecitabine; Drug: docetaxel

INTERVENTIONS:
Drug: capecitabine — Participants received capecitabine according to individualized physician-prescribed regimen.
Drug: docetaxel — Participants received docetaxel according to individualized physician-prescribed regimens.

SUMMARY:
This multicenter observational study will evaluate the efficacy and safety of Xeloda (capecitabine) in combination with docetaxel in first-line therapy in participants with HER2-negative metastatic breast cancer. Participants will be followed for approximately 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* HER2-negative metastatic breast cancer
* Participants initiated on first-line therapy with Xeloda and docetaxel in accordance with the Summary of Product Characteristics; participants who started treatment with Xeloda and docetaxel no more than 3 months before enrollment in this study are also eligible

Exclusion Criteria:

* Contraindications to Xeloda treatment according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HER2-negative metastatic breast cancer initiated on first-line therapy with Xeloda in combination with docetaxel
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Hungary (11):
  - Budapest
  - Debrecen
  - Gyula
  - Kaposvár
  - Kecskemét
  - Miskolc
  - Nyíregyháza
  - Szeged
  - Szombathely
  - Veszprém
  - Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 participants were enrolled in the study and included in safety assessments. 45 participants were included in other assessments.
Period: Overall Study
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Started | 46
Evaluable Participants | 45
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were female.
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.58 (11.359)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The time from enrollment until disease progression, assessed as the time to tumor progression, as evaluated by regular examinations per routine clinical practice, or death from any cause.
Time Frame: approximately 2 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
months | 9.89 (2.97)

2. Secondary Outcome: Time to Treatment Failure
Description: The time from enrollment to discontinuation of any drug of the treatment combination.
Time Frame: approximately 2 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
months | 4.64 (5.14)

3. Secondary Outcome: Overall Response Rate
Description: The percentage of participants with complete or partial remission, based on evaluation of tumor responses assessed at regular examinations per routine clinical practice.
Time Frame: approximately 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
percentage of participants | 28.9

4. Secondary Outcome: Clinical Benefit Rate
Description: The percentage of participants with an overall response (complete or partial remission) or with stable disease.
Time Frame: approximately 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
percentage of participants | 73.3

5. Secondary Outcome: Duration of Treatment With Xeloda
Time Frame: approximately 2 years
Measure: Mean (Standard Deviation); unit: treatment cycle
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
treatment cycle | 6.24 (4.80)

6. Secondary Outcome: Percentage of Capecitabine Dose Modifications
Time Frame: approximately 2 years
Measure: Number; unit: percentage of doses
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 45
percentage of doses | 44.4

7. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: approximately 2 years
Population: 46 participants enrolled in the study were evaluable with regards to tolerability; however, 1 participant did not meet the eligibility criteria, was excluded from the efficacy analyses, but was included in the safety analyses.
Measure: Number; unit: participants
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Number analyzed (Participants) | 46
participants | 33

ADVERSE EVENTS:
Arm/Group | Participants Receiving Capecitabine/Docetaxel
Serious Adverse Events (participants affected / at risk) | 8/46
Other Adverse Events (participants affected / at risk) | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving Capecitabine/Docetaxel (N=46)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Disease Progression (General disorders) | 3 (3)
Mucositis (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving Capecitabine/Docetaxel (N=46)
Neutropenia (Blood and lymphatic system disorders) | 10 (14)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Mucositis (General disorders) | 4 (4)
Palmoplantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.